CLINICAL TRIAL: NCT03414177
Title: Telehealth Enhanced Asthma Management
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207015
Record Dates: First submitted 2018-01-09; First posted 2018-01-29 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: Telemedicine; Clinical follow up visits
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: One group will receive asthma follow up care via telemedicine at a remote clinical sites. The second group will receive in-person asthma follow-up care at a specialty clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group (Active Comparator): Telemedicine participants will have asthma subspecialty follow-up visits conducted via real-time audio and video conferencing in conjunction with electronic examination peripherals and remote pulmonary function testing (PFT). Participants will receive a survey link to complete an electronic survey to assess Asthma Control Test (ACT) score, healthcare utilization, and satisfaction.
  Interventions: Other: Asthma Subspecialty Follow-up Visits
- In-Person Group (Active Comparator): In-Person participants will have asthma subspecialty follow-up visits at a subspecialty clinic. They will receive pulmonary function testing (PFT). Participants will receive a survey link to complete an electronic survey to assess Asthma Control Test (ACT) score, healthcare utilization, and satisfaction.
  Interventions: Other: Asthma Subspecialty Follow-up Visits

INTERVENTIONS:
Other: Asthma Subspecialty Follow-up Visits — Pediatric patients with persistent asthma will be recruited to compare outcomes among patients with follow-up visits managed via telemedicine vs. in-person visits.

SUMMARY:
This study will conduct a 12-month randomized trial with 48 pediatric patients (aged 6-18 years) with persistent asthma to compare outcomes among patients with follow-up visits managed via telemedicine (TM) vs. in-person (IP) visits.

DETAILED DESCRIPTION:
The overarching hypothesis is that utilization of TM for asthma follow-up will result in improved clinical outcomes such as Asthma Control Test (ACT) scores, lung function and medication adherence compared to participants receiving IP follow-up care. The Investigator also hypothesize that TM follow-up will result in higher caregiver satisfaction because families will be able to receive quality subspecialty care in their community (TM) compared to those who travel a distance to receive care (IP).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥6- and ≤18 years
2. persistent asthma as defined by national guidelines standards
3. receives care at an ACH asthma subspecialty clinic
4. reside ≤1.5 hour drive from Jonesboro, Springdale, Texarkana, or Fort Smith, AR

Exclusion Criteria:

1. Significant underlying respiratory disease other than asthma, such as cystic fibrosis
2. significant co-morbid conditions, such as individuals with developmental or physical impairments that could interfere with the ability to communicate via interactive video
3. current smoker
4. severe asthma exacerbation requiring intubation in the past 12 months
5. no access to a smartphone or internet

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Mean difference in ACT score at the final assessment (12 months) after adjusting for baseline | At baseline and 12 months
  ACT is used for symptoms monitoring as per guidelines and has been identified as an appropriate asthma control composite score in clinical research.

SECONDARY OUTCOMES:
Routine Follow up Asthma Visit | At baseline, 4 months, 8 months, 12 months
  Physical examination to assess current asthma problems, symptoms, medication and the child's overall health.
Lung Function via Spirometry | Baseline and 12 months
  Spirometry
Airway Inflammation via Spirometry | Baseline and 12 months
  Spirometry
Healthcare Utilization | At baseline, 4 months, 8 months, 12 months
  Patient report of the number of acute exacerbation in the past 12 months resulting in hospitalizations, emergency room or sick visits or steroid use.
Medication Adherence | At baseline, 4 months, 8 months, 12 months
  Adherence will be defined as receiving ≥3 controller medication refills/6 months or achieving an Asthma Medication Ratio (AMR) of ≥0.5 based on national asthma guidelines.
Rescue Medication Use | At baseline, 4 months, 8 months, 12 months
  Assessment of rescue medication use by caregiver report.
Clinic Visit Attendance Rate | At baseline, 4 months, 8 months, 12 months
  Participant clinic attendance / Completion rate for Telemedicine and In-Person group.
Visit Satisfaction | At baseline, 4 months, 8 months, 12 months
  Participant report of satisfaction with asthma follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, MD, Principal Investigator — Arkansas Children's Research Institute
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No